CLINICAL TRIAL: NCT00175812
Title: Differentiation Induction Therapy for Acute Myelogenous Leukemia
Brief Title: Differentiation Induction in Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Øystein Bruserud, Professor, University of Bergen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK-Vestnr21503
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Acute myelogenous leukemia; Differentiation; All trans retinoic acid; Valproic acid; Theophyllamin
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Tretinoin; Valproic Acid; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATRA plus valproic acid plus theophyllin (Experimental): ATRA for 14 days, continuous treatment with valproic acid and theophyllin
  Interventions: Drug: all-trans retinoic acid (ATRA); Drug: Valproic acid; Drug: Theophyllin

INTERVENTIONS:
Drug: all-trans retinoic acid (ATRA) — All-trans retinoic acid 22.5 mg/square meter twice daily days 1-14
Drug: Valproic acid — Valproic acid, highest dose without side effects from day 3 until progression
Drug: Theophyllin — Theophyllin, targetted serum level 50-100 from day 3 until progression

SUMMARY:
Hypothesis: Differentiation induction therapy in acute myelogenous leukemia (AML) can be used to achieve disease control and stabilize peripheral blood counts in patients with acute myelogenous leukemia.

Adult patients (<18 years of age) who can be included: Elderly patients (>60 years of age) with newly diagnosed AML who cannot achieve standard chemotherapy, patients with relapsed or resistant AML. Patients with relapsed or resistant AML who cannot receive intensive chemotherapy.

Treatment: Patients will be treated with all-trans retinoic acid (oral administration), valproic acid (7 days intravenous administration and later oral administration)and theophyllamine (7 days intravenous administration and later oral administration). Duration of treatment at least 2 months or until disease progression. Maximal duration of treatment 2 years.

Followup: Clinical evaluation, peripheral blood samples, bone marrow samples.

DETAILED DESCRIPTION:
Patients to be included:

1. Elderly patients above 60 years of age with newly diagnosed acute myelogenous leukemia (AML) who cannot receive conventional intensive chemotherapy.
2. Adult patients of any age (> 18 years of age)with relapsed or resistant AML who cannot receive conventional intensive chemotherapy or allogeneic stem cell transplantation.

We plan to include at least 20 patients, but if possible 30 patients during a 3 years period. The first patient was included November 2004.

Treatment:

All-trans retinoic acid (ATRA) administered orally 22.5 mg/m2 twice daily for 14 days, repeated every third month.

Valproic acid started on day 3 of ATRA therapy, the first week as intravenous administration and later oral administration.

Theophyllamine started on day 3 of ATRA therapy, the first week as intravenous administration and later oral administration.

Duration of treatment at least 2 months unless side effects,until disease progression or an overall duration of treatment of 2 years.

Supportive therapy according to the hospitals general guidelines.

Followup:

The first week treatment in hospital. Later out-patient treatment with regular controls including clinical examination, peripheral blood parameters (including serum valproic acid and theophyllamin levels), bone marrow samples.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed acute myelogenous leukemia (AML)
* Patients above 60 years of age
* Patients who cannot receive conventional chemotherapy
* Patients with relapsed or refractory AML independent of age

Exclusion Criteria:

* Chronic myelogenous leukemia in blast phase
* Intolerance to the study drugs
* Serious liver disease
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Survival | 2008

SECONDARY OUTCOMES:
Disease stabilisation | 2008
Disease complications | 2008
Side effects of therapy | 2008

CONTACTS AND LOCATIONS:
Overall Officials: Oystein Bruserud, MD, Principal Investigator — University of Bergen
Locations (1):
- Haukeland University Hospital, University of Bergen, Bergen, Norway

REFERENCES:
- [Result] Ryningen A, Stapnes C, Lassalle P, Corbascio M, Gjertsen BT, Bruserud O. A subset of patients with high-risk acute myelogenous leukemia shows improved peripheral blood cell counts when treated with the combination of valproic acid, theophylline and all-trans retinoic acid. Leuk Res. 2009 Jun;33(6):779-87. doi: 10.1016/j.leukres.2008.10.005. Epub 2008 Nov 12. PMID 19007987
- [Result] Ryningen A, Stapnes C, Paulsen K, Lassalle P, Gjertsen BT, Bruserud O. In vivo biological effects of ATRA in the treatment of AML. Expert Opin Investig Drugs. 2008 Nov;17(11):1623-33. doi: 10.1517/13543784.17.11.1623. PMID 18922099
- [Derived] Haaland I, Hjelle SM, Reikvam H, Sulen A, Ryningen A, McCormack E, Bruserud O, Gjertsen BT. p53 Protein Isoform Profiles in AML: Correlation with Distinct Differentiation Stages and Response to Epigenetic Differentiation Therapy. Cells. 2021 Apr 7;10(4):833. doi: 10.3390/cells10040833. PMID 33917201
- [Derived] Reikvam H, Hovland R, Forthun RB, Erdal S, Gjertsen BT, Fredly H, Bruserud O. Disease-stabilizing treatment based on all-trans retinoic acid and valproic acid in acute myeloid leukemia - identification of responders by gene expression profiling of pretreatment leukemic cells. BMC Cancer. 2017 Sep 6;17(1):630. doi: 10.1186/s12885-017-3620-y. PMID 28877686
- [Derived] Skavland J, Jorgensen KM, Hadziavdic K, Hovland R, Jonassen I, Bruserud O, Gjertsen BT. Specific cellular signal-transduction responses to in vivo combination therapy with ATRA, valproic acid and theophylline in acute myeloid leukemia. Blood Cancer J. 2011 Feb;1(2):e4. doi: 10.1038/bcj.2011.2. Epub 2011 Feb 11. PMID 22829110